CLINICAL TRIAL: NCT01777100
Title: Phase IV Study of Postoperative Analgesic Efficacy and Safety of Anesthesia Induction With Single Dose Sufentanil for Open Abdominal Surgery Under Continuous Remifentanil Anesthesia Versus Total Intravenous Remifentanil Anesthesia
Brief Title: Sufentanil for Anesthesia Induction in Continuous Remifentanil Anesthesia
Acronym: SAIRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernanda Bono Fukushima, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNESP
Record Dates: First submitted 2012-07-02; First posted 2013-01-28 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Patient controlled analgesia; Hyperalgesia; Remifentanil; Sufentanil; Morphine; Abdominal surgery; Safety
MeSH Terms: conditions — Pain, Postoperative; Hyperalgesia | interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sufentanil (Experimental): Anesthetic induction with IV sufentanil at 0.5 mcg.kg-1 and analgesic maintenance with IV remifentanil at 0.1 to 0.3 mcg.kg-1.min-1 on demand target-controlled infusion
  Interventions: Drug: Sufentanil
- remifentanil (No Intervention): Anesthetic induction with target-controlled infusion IV remifentanil at 0.5 mcg.kg-1.min-1 in 5 minutes followed by analgesic maintenance on demand of IV target-controlled infusion remifentanil at 0.1 to 0.3 mcg.kg-1.min-1.

INTERVENTIONS:
Drug: Sufentanil — Sufentanil 0.5 mcg.kg-1 at anesthesia induction (single dose)
  Other Names: CAS number 56030-54-7; ATC code N01AH03; PubChem CID 41693; DrugBank DB00708; ChemSpider 38043; UNII AFE2YW0IIZ; KEGG D05938 Yes; ChEBI CHEBI:9316; ChEMBL CHEMBL658; Formula C22H30N2O2S
  Arms: sufentanil

SUMMARY:
The appropriate management of postoperative pain is recognized as an important clinical challenge with implications beyond humanitarian issues. Evidence shows that effective postoperative analgesia is associated with physiological benefits to the patient, shortened length of hospital stay and lower rates of in-hospital complications, such as pneumonia, delirium and persistent pain after surgery. However, despite the availability of several analgesic drugs and strategies the prevention and treatment of postoperative pain is often suboptimal. Remifentanil is a potent short acting opioid commonly used in continuous infusion for anesthesia for several surgical procedures. Remifentanil has been extensively advocated as a means to provide quick patient awakening in the immediate postoperative period with a very low risk of respiratory depression. Yet it does not provide residual analgesia and postoperative pain is a major concern. In order to overcome this limitation, practicing anesthesiologists frequently give patients a single dose of Sufentanil, a long acting opioid, during the induction of anesthesia where Remifentanil will be used in continuous infusion. However the effectiveness of this strategy still lacks evidence from controlled clinical trials.

DETAILED DESCRIPTION:
We propose the current randomized clinical trial to assess the analgesic effectiveness of Sufentanil administered as a single dose during the induction of anesthesia for the management of postoperative pain in patients undergoing open abdominal surgery performed with continuous infusion of Remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* Physical status (American Society of Anesthesiologists) 1, 2 or 3
* Age 18 years and older
* Patients selected for open Abdominal surgery under general total intravenous anesthesia

Exclusion Criteria:

* Physical status (American Society of Anesthesiologists) 4
* Patients undergoing other anesthesia technic (subarachnoid, epidural, nerve block, etc)
* History of anaphylactic reaction after use of tramadol, dipyrone, propofol, rocuronium, dexamethasone, sufentanil, remifentanil or morphine
* Chronic uso of drugs that are associated with major increases in the activity of P450 isozymes (Carbamazepine, phenobarbital, rifampin, tobacco, phenytoin, Hypericum perforatum)
* Previous History of Drug addiction
* alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption through patient controlled analgesia pump | 24 hours after surgery

SECONDARY OUTCOMES:
Morphine consumption through patient controlled analgesia pump | 15 minutes after arrival at post-anesthesia care unit
Morphine consumption through patient controlled analgesia pump | 30 minutes after arrival at post-anesthesia care unit
Morphine consumption through patient controlled analgesia pump | 60 minutes after arrival at post-anesthesia care unit
Morphine consumption through patient controlled analgesia pump | 12 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda B Fukushima, MD PhD, Principal Investigator — UPECLIN HC FM Botucatu Unesp
Locations (1):
- Faculdade de Medicina de Botucatu, Botucatu, São Paulo, Brazil